CLINICAL TRIAL: NCT04806230
Title: Serum Concentrations of Antidepressant Drugs in Pregnant Women - a Naturalistic Study
Acronym: PAPA
Status: Completed | Type: Observational
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Erik Nilzén, MD, Linkoeping University
Other Study IDs: PAPA123
Record Dates: First submitted 2021-03-15; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Pharmacokinetics; Antidepressive Agents; Pregnancy
Keywords: Pharmacokinetics; antidepressants; pregnancy
MeSH Terms: interventions — Sertraline; Mirtazapine; Venlafaxine Hydrochloride; Citalopram; Escitalopram

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observed
  Interventions: Drug: sertraline, mirtazapine, venlafaxine, citalopram, escitalopram

INTERVENTIONS:
Drug: sertraline, mirtazapine, venlafaxine, citalopram, escitalopram — Naturalistic treatment

SUMMARY:
The study was a prospective naturalistic PK study of five frequently used antidepressant drugs in pregnant women; citalopram (CIT), escitalopram (ECIT), sertraline (SERT), mirtazapine (MIRT) and venlafaxine VEN) and their major metabolites (Table 1). After signing informed consent pregnant women with ongoing antidepressant treatment, regardless of indication, were recruited at nine antenatal care centers in mid- and small cities and villages in the Southeast Sweden between April 2011 and September 2013.

DETAILED DESCRIPTION:
Serum samples for the antidepressant drug and metabolite(s) concentrations, albumin and creatinine were collected at the first prenatal appointment and at gestational week 15, 20, 25, 35 and at partus. The time interval between drug intake and sampling was registered in all cases. At partus, a serum samples from the umbilical cord was collected drug concentration was assessed. At the first prenatal appointment a blood sample for analyzing the CYP2D6 and CYP2C19 genotype was also collected. All drug concentration analysis were executed post hoc, after last partus, whereas physiological parameters were part of normal routine sampling. Concomitant medication, weight changes and smoking habits were registered throughout the pregnancies.

Our main findings were that dose corrected serum concentrations of neither sertralin nor citalopram changed during the pregnancy. In addition, concentrations of escitalopram and venlafaxine and their metabolites appeared to be stable throughout pregnancy, even though a linear mixed models statistic calculation could not be done due small number of samples.

Results from previous research on sertraline PK during pregnancy are inconclusive. Two studies suggested decreased levels (Freeman, Sit 2), while one study indicated increased levels (Westin). Previous studies, except for Westin's are, however, limited by small sample sizes (six and eight) and a substantial inter-individual variance.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy
* Ongoing treatment with one of the five studied antidepressants.

Exclusion Criteria:

• None

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: At inclusion, median age (min-max) was 31 years (21-42) and median BMI was 25.6 (18.9-47.0)
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2011-04-01 (Actual); Primary Completion 2013-09-30 (Actual); Study Completion 2013-09-30 (Actual)

PRIMARY OUTCOMES:
Serum concentrations of drugs and metabolites | 9 months
  levels of parent compound and metabolites in serum

CONTACTS AND LOCATIONS:
Locations (1):
- Linköping University, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No